CLINICAL TRIAL: NCT01756625
Title: Factors Impacting on Efficacy and Compliance to Cetuximab Treatment in First Line WT KRAS Metastatic Colorectal Cancer
Brief Title: PREMIUM, Observational Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr.Laurent Mineur (Other)
Collaborators: Merck Serono International SA (Industry); BESPIM, CHU Nîmes (data analysis) (Unknown)
Responsible Party: Sponsor-Investigator, Dr.Laurent Mineur, Oncologist, Institut Sainte Catherine
Organization: Institut Sainte Catherine (Other)
Other Study IDs: PREMIUM
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: First Line WT KRAS mCRC
Keywords: cetuximab; nicotine; magnesium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First line WT KRAS mCRC

SUMMARY:
PREMIUM is an observational pharmaco-epidemiologic, transversal, multi-centric, prospective cohort study and with independent investigators. The purpose is to compare PFS in real life with PFS clinical trials and to determine factors impacting efficacy and compliance to cetuximab treatment in first line K-ras wild-type (wt) metastatic colorectal cancer.

DETAILED DESCRIPTION:
Retrospective studies have shown the influence of some factors on the efficacy of treatment with cetuximab (nicotine, magnesium etc..). No randomized study has compared the mode of administration of weekly and biweekly cetuximab. What are the factors influencing patient compliance? Adverse events, the relation between doctor and patient. PREMIUM will attempt to explore and assess the variables associated with efficacy and compliance to treatment and study practices in France for clinical management.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old diagnosed with mCRC
* patients naïve for CT excepted for adjuvant setting or trated max 2 cycles CT in first line mCRC with or without cetuximab
* all patients receiving cetuximab in first line treatment associated or not with CT
* patients relapsed < 6 months after an adjuvant therapy

Exclusion Criteria:

* patients participating to clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from private and public centers
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
To compare PFS rate at 1 year with PFS in clinical studies (ITT and subgroup analysis) | 3 years

SECONDARY OUTCOMES:
ORR at 1 year (ITT and subgroup analysis) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Sainte-Catherine, Avignon, Vaucluse, France

REFERENCES:
- [Derived] Mineur L, Francois E, Plassot C, Phelip JM, Miglianico L, Dourthe LM, Bonichon N, Moreau L, Guimbaud R, Smith D, Achille E, Herve R, Bons JM, Remy S, Faroux R, Villing AL, Mahamat A, Rabbia I, Soulie P, Baumgaertner I, Mathe N, Vazquez L, Boustany R. PREMIUM: A French prospective multicenter observational study of factors impacting on efficacy and compliance to cetuximab treatment in first-line KRAS wild-type metastatic colorectal cancer. PLoS One. 2020 Dec 21;15(12):e0243997. doi: 10.1371/journal.pone.0243997. eCollection 2020. PMID 33347495